CLINICAL TRIAL: NCT06966180
Title: Development and Evaluation of the Effectiveness of an Alcohol Intervention Program for Adults on Probation: A Randomized Controlled Trial
Brief Title: Development and Effectiveness of an Alcohol Intervention Program for Adults Under Probation
Acronym: PROB-AIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mine Pazarcikci (Other)
Responsible Party: Sponsor-Investigator, Mine Pazarcikci, PhD, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-AIP-2025; 22-10.1T/32 (Registry Identifier: Medical Research Ethics Committee of Ege University)
Record Dates: First submitted 2025-05-03; First posted 2025-05-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder; Problem Drinking; Psychosocial Intervention
Keywords: Alcohol Use; Alcohol Intervention; Criminal Justice System; Probation; Psychosocial Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention or the control group.
Who Masked: Participant
Masking Description: Single-blind design; participants were not informed about group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol Intervention Program (AIP) (Experimental): Participants received a structured Alcohol Intervention Program (AIP) consisting of six bi-weekly group sessions. The program was based on motivational interviewing and cognitive-behavioral strategies and aimed to reduce alcohol use and related problems while increasing motivation to change.
  Interventions: Behavioral: Alcohol Intervention Program (AIP)
- Probation Only (No Psychosocial Intervention) (No Intervention): Participants in this group did not receive any intervention program during the study period. They continued with standard probation supervision without any additional psychosocial intervention components.

INTERVENTIONS:
Behavioral: Alcohol Intervention Program (AIP) — A brief behavioral intervention consisting of six bi-weekly group sessions based on motivational interviewing and cognitive-behavioral strategies. The aim was to reduce alcohol use and related problems and increase motivation to change.
  Arms: Alcohol Intervention Program (AIP)

SUMMARY:
The aim of this study is to develop and evaluate the effectiveness of an alcohol-specific intervention program for adult individuals on probation who have problems related to alcohol use. The study was designed as a single-blind randomized controlled trial and was conducted at the Izmir Probation Directorate with a total of 115 participants, 58 in the intervention group and 57 in the control group. When comparing the results between the intervention and control groups, the Alcohol Intervention Program-which consisted of six structured sessions-was found to be effective in reducing participants' alcohol consumption and related problems, while also increasing their motivation for change. This research is significant as it represents the first intervention program developed specifically for alcohol use within the probation system. While existing interventions in both Turkey and abroad often focus on individuals who use illicit substances, alcohol-related problems are frequently overlooked. The results of this study aim to meet that systemic need. The Alcohol Intervention Program developed here can be integrated into routine practices within the scope of educational improvement programs in the probation system.

DETAILED DESCRIPTION:
This study aimed to develop and evaluate the effectiveness of a structured Alcohol Intervention Program (AIP) for adults under probation who experience alcohol-related problems. The research was designed as a single-blind randomized controlled trial and was conducted at the Izmir Probation Directorate in Turkey between June and November 2023. A total of 115 participants were recruited and randomly assigned to an intervention group (n = 58) and a control group (n = 57). The intervention group received a structured program consisting of six bi-weekly sessions based on motivational interviewing and cognitive-behavioral strategies. No intervention program was administered to the control group. Standardized self-report tools, including the Alcohol Use Disorders Identification Test (AUDIT), the Michigan Alcoholism Screening Test (MAST), and the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES), were administered as pre- and post-tests. Statistical analysis included paired-samples t-tests, independent-samples t-tests, ANOVA, chi-square, and regression analysis. The results showed that participants in the intervention group demonstrated a significant reduction in alcohol use and related problems, as well as a significant increase in motivation to change, compared to the control group. The study demonstrates that the AIP is effective in supporting rehabilitation within the probation system and highlights the need for structured, alcohol-specific programs in this context. This research is significant in that it represents the first intervention program developed specifically for alcohol use within the probation system in Turkey. The findings suggest that the program can be integrated into existing probation practices and adapted to other contexts with similar needs. This study helps fill an important gap in the system and provides a foundation for future large-scale implementation research.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Willingness to participate in the study (providing informed consent)
* Being literate
* Being under probation supervision and experiencing problems related to alcohol use, such as:
* Problematic alcohol consumption
* Endangering traffic safety due to alcohol use
* Committing an offense under the influence of alcohol

Exclusion Criteria:

* Having a psychotic disorder
* Use of any psychoactive or addictive substances other than alcohol
* Currently receiving treatment for alcohol-related problems voluntarily and outside the scope of probation supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Reduction in Alcohol Use (AUDIT Score) | From baseline to study completion (Week 12, immediately after completion of the 6-session program)
  The primary outcome was the change in participants' alcohol consumption, measured by the Alcohol Use Disorders Identification Test (AUDIT). The AUDIT consists of 10 items with a total score range of 0 to 40. Higher scores reflect more severe alcohol use. The effectiveness of the Alcohol Intervention Program (AIP) was evaluated by comparing AUDIT scores at baseline and at the end of the study (Week 12, immediately after the last session). A significant reduction in scores indicated decreased alcohol use and fewer alcohol-related problems.

SECONDARY OUTCOMES:
Reduction in Alcohol-Related Problems (MAST Score) | From baseline to study completion (Week 12, immediately after completion of the 6-session program)
  This secondary outcome assessed changes in alcohol-related problems using the Michigan Alcoholism Screening Test (MAST). The MAST consists of 25 items with a total score range of 0 to 53. Higher scores indicate alcohol-related problems and impairments in social functioning. Scores at baseline and at the end of the study (Week 12) were compared, and reductions indicated improvements in alcohol-related problems.
Increase in Motivation to Change (SOCRATES Score) | From baseline to study completion (Week 12, immediately after completion of the 6-session program)
  This outcome measured participants' motivation to change their alcohol use behaviors using the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES). The version used in this study included 19 items with a total score range of 19 to 95. Higher scores indicated greater readiness for change and stronger motivation to reduce alcohol use. Scores at baseline and at the end of the study (Week 12) were compared, and an increase in scores reflected a rise in participants' motivation to change.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Pazarcıkcı, PhD, Principal Investigator — Ege University
Locations (1):
- İzmir Probation Directorate, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No